CLINICAL TRIAL: NCT00004889
Title: Phase II Study of Rituximab (Rituxan, Mabthera) in Waldenstrom's Macroglobulinemia
Brief Title: Rituximab in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Christos Emmanouilides, MD / Principal Investigator, UCLA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067565; UCLA-9909016; NCI-G00-1709
Record Dates: First submitted 2000-03-07; First posted 2004-02-12 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituxan (Experimental): 375 mg/m2 given as an intravenous (IV) infusion once weekly for four doses (days 1, 8, 15, and 22). For purposes of this study 4 weekly courses will constitute one cycle of therapy.
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — 375 mg/m2 given as an intravenous (IV) infusion once weekly for four doses (days 1, 8, 15, and 22). For purposes of this study 4 weekly courses will constitute one cycle of therapy.
  Other Names: Rituxan

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab in treating patients who have Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response, time to treatment failure, and toxicity in patients with Waldenstrom's macroglobulinemia treated with rituximab. II. Correlate expression and changes in expression of CD20 on patient plasma cells and B-cells with clinical responses.

OUTLINE: This is a multicenter study. Patients receive rituximab IV weekly for 4 weeks. Treatment may be repeated 2 months later in patients with stable disease, partial response, or complete response. Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 12-25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Waldenstrom's Macroglobulinemia requiring therapy who have received no more than 2 prior courses of therapy; previously untreated patients with slowly progressive WM if the patient can reasonably be expected to not require chemotherapy or steroid therapy for 90 days
* CD20 positive tumor cells
* Presence of monoclonal paraprotein
* Minimum IgM level > 2 times the upper limit of normal
* Adequate organ function: ANC>1000/uL; PLT > 25000/uL; serum creatinine < 2.5; serum total bilirubin and SGOT < 2.5 times the upper limit of normal
* 18 years and older
* Life expectancy of 6 months or greater
* ECOG performance status of 0-2
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for 6 months after completion of treatment

Exclusion Criteria:

* Chemotherapy, steroid therapy, or radiation therapy within 30 days of study entry
* Patients who are pregnant
* Serious co-morbid disease
* Uncontrolled bacterial, fungal, or viral infection
* Active second malignancy
* Individuals who cannot provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1999-12; Primary Completion 2002-01 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Response (delay in disease progression or timing of disease progression) | 24 weeks
  Define objective response (delay in disease progression or timing of disease progression), time to treatment failure, and toxicity for single agent Rituxan therapy in Waldenstrom's macroglobulinemia patients

SECONDARY OUTCOMES:
Expression of CD20 | 24 weeks
  To correlate expression and changes in expression of CD20 on waldenstrom's macroglobulinemia patient plasma cells and B-cells with clinical responses.

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (8):
- United States (7):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Cross Cancer Institute, Edmonton, Alberta, Canada